CLINICAL TRIAL: NCT04453423
Title: A Study of the Effect of Anlotinib, Pemetrexed or the Combination As Maintenance Therapy for Patients With Non-Squamous Non-Small Cell Lung Cancer.
Brief Title: Combination Chemotherapy With or Without Anlotinib in the Maintenance Treatment of Non-Squamous Non-Small Cell Lung Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AN001
Record Dates: First submitted 2020-06-27; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Non-squamous Non-small-cell Lung Cancer
MeSH Terms: interventions — anlotinib; Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- First-line Treatment (Other)
  Interventions: Drug: Anlotinib + Pemetrexed+Carboplatin
- Maintenance Treatment A (Experimental)
  Interventions: Drug: Pemetrexed
- Maintenance Treatment B (Experimental)
  Interventions: Drug: Anlotinib + Pemetrexed
- Maintenance Treatment C (Experimental)
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib + Pemetrexed+Carboplatin — Anlotinib: 12mg, QD, PO, d1-14, 21 days per cycle
  Carboplatin: AUC 5 on day 1 of 21 days per cycle
  Pemetrexed: 500mg/m2 iv on day 1 of 21 days per cycle
  Arms: First-line Treatment
Drug: Pemetrexed — 500mg/m2 iv on day 1 of 21 days per cycle(maintenance phase)
  Arms: Maintenance Treatment A
Drug: Anlotinib + Pemetrexed — Anlotinib:12mg, QD, PO, d1-14, 21 days per cycle(maintenance phase)
  Pemetrexed:500mg/m2 iv on day 1 of 21 days per cycle(maintenance phase)
  Arms: Maintenance Treatment B
Drug: Anlotinib — 12mg, QD, PO, d1-14, 21 days per cycle(maintenance phase)
  Arms: Maintenance Treatment C

SUMMARY:
This study will compare maintenance therapy with anlotinib plus pemetrexed versus pemetrexed or anlotinib alone, in patients with Non-squamous Non-small cell lung cancer who have not progressed during first-line therapy with anlotinib + pemetrexed + carboplatin. The primary endpoint of the study is progression-free survival (PFS); the secondary endpoints are disease control rate (DCR), objective response rate (ORR) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 75, ECOG PS: 0~1, estimated survival duration more than 3 months;
2. Subjects with histologically or cytologically confirmed locally advanced and/or advanced Non-squamous NSCLC;
3. Signed and dated informed consent;
4. adequate hematological, liver and renal function

Exclusion Criteria:

1. prior chemotherapy or treatment with another systemic anti-cancer agent
2. malignancies other than NSCLC within 5 years prior to randomization, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer or DCIS
3. evidence of tumor invading major blood vessels
4. current or recent use of aspirin (>325mg/day) or full-dose anticoagulants or thrombolytic agents for therapeutic purposes
5. history of haemoptysis >/=grade 2
6. clinically significant cardiovascular disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 6 months
  PFS is defined as the time from the date of treatment to the first date of disease progression or death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 12 months)
  Treatment response are defined as complete response (CR), partial response (PR), stable disease (SD) and progression disease (PD) according to Response Evaluation Criteria in Solid Tumor (RECISIT criteria, version 1.1). The percentage of patients who achieved CR and PR was defined as objective response rate (ORR).
Disease control rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 12 months)
  Treatment response are defined as complete response (CR), partial response (PR), stable disease (SD) and progression disease (PD) according to Response Evaluation Criteria in Solid Tumor (RECISIT criteria, version 1.1) and the percentage of patients who achieved CR, PR and SD was defined as disease control rate (DCR).
Overall Survival (OS) | 12 months
  OS is calculated from diagnosis to death or last follow-up time.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Until 30 day safety follow-up visit
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability